CLINICAL TRIAL: NCT04751539
Title: A Randomized, Double-Blind, Placebo-Controlled Dose-Escalation Study in Healthy Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AND017 Following Oral Single and Multiple Dose Administration
Brief Title: A Dose-escalation Study of AND017 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kind Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BB-AND017AU001
Record Dates: First submitted 2021-01-28; First posted 2021-02-12 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AND017 single dose escalation (Experimental): Subjects will be administrated with single dose of AND017 capsule from 1 mg to 50 mg during Part A.
  Interventions: Drug: AND017 single dose
- AND017 repeated dose escalation (Placebo Comparator): Subjects will be administrated with repeated dose of AND017 from 4 mg to 30 mg for 10 consecutive days during Part B.
  Interventions: Drug: AND017 multiple dose
- Placebo (Placebo Comparator): Placebo administrated once on Day 1 in Part A or daily from Day 1 to Day 10 in Part B
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AND017 single dose — AND017 administrated as oral single-dose on Day 1 in Part A
  Arms: AND017 single dose escalation
Drug: AND017 multiple dose — AND017 administrated once daily from Day 1 to Day 10 in Part B
  Arms: AND017 repeated dose escalation
Drug: Placebo — Placebo administrated once on Day 1 in Part A or daily from Day 1 to Day 10 in Part B
  Arms: Placebo

SUMMARY:
This is a phase I, randomized, double-blind, placebo-controlled, dose-escalation study in healthy subjects to evaluate safety, tolerability, PKs and PDs of AND017 following oral single and multiple dose administration.

ELIGIBILITY:
Inclusion Criteria:

1. BMI within 18.0-30.0 kg/m2 (inclusive)
2. Blood Pressure (BP) and 12-lead electrocardiogram (ECG) showing no clinically significant abnormalities during screening;
3. No clinically significant abnormal values in physical examination, clinical laboratory tests, liver function or kidney function;

Exclusion Criteria:

1. Current or chronic history of liver disease or known hepatic or biliary abnormalities, including but not limited to ALT, alkaline phosphatase and bilirubin >1.5xULN (isolated bilirubin>1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%);
2. Subjects with Hb: male <120 g/L or >160 g/L, female <110 g/L or >150 g/L;
3. Subjects with any abnormalities of hematology during screening: Mean corpuscular volume (MCV), platelet count, serum iron, ferritin;
4. Subjects with a history of medical treatment or disease likely to increase the risk of bleeding or disturbance of blood coagulation;
5. History of deep vein thrombosis, stoke, transient ischemic attack, pulmonary embolism or other thrombosis-related condition within the last five years;
6. History of myocardial infarction, heart failure or acute coronary syndrome;
7. Evidence of active peptic, duodenal or esophageal ulcer disease at screening;
8. History of pulmonary artery hypertension;
9. History of sensitivity to heparin or heparin-induced thrombocytopenia;
10. Subjects with major illness or surgery within past 3 months prior to screening, or planned surgery during study;
11. Known or suspected history of drug abuse within the past 5 years or presence of drug abuse within 3 months before study;
12. Donated blood >400 mL or significant blood loss equivalent to 400 mL or received blood transfusion within 3months of screening; or donated blood >200 mL or significant blood loss equivalent to 200 mL within 1 month prior to screening.
13. Participation in any clinical study with an investigational drug, biologic or device within 4 weeks or 5 times the half-life of the specific drug/biologics (whichever is longer), prior to dosing;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Safety evaluations | 17 Days
  Incidents of AE and abnormal laboratory tests

SECONDARY OUTCOMES:
Plasma Cmax of AND017 | 1 day
  The plasma Cmax of AND017 by single dose administration
Plasma Tmax of AND017 | 1 day and 10 days
  The plasma Tmax of AND017 after single dose administration on D1 and multiple doses for 10 consecutive days on D10
Plasma t1/2 of AND017 | 1 day and 10 days
  The plasma T1/2 of AND017 after single dose administration on D1 and multiple doses for 10 consecutive days on D10
Plasma AUC of AND017 | 1 day and 10 days
  The plasma AUCs of AND017 after single dose administration on D1 and multiple doses for 10 consecutive days on D10
Plasma CL/F of AND017 | 1 day
  The plasma CL/F of AND017 after single dose administration
Plasma Vz/F of AND017 | 1 day
  The plasma Vz/F of AND017 after single dose administration
Plasma MRT of AND017 | 1 day
  The plasma MRT of AND017 after single dose administration
Plasma λz of AND017 | 1 day
  The plasma λz of AND017 after single dose administration
Plasma %AUCex of AND017 | 1 day
  The plasma %AUCex of AND017 after single dose administration
Plasma Css,min of AND017 | 10 days
  The plasma Css,min of AND017 by multiple administration for 10 consecutive days
Plasma Css,max of AND017 | 10 days
  The plasma Css,max of AND017 by multiple administration for 10 consecutive days
Plasma Css,avg of AND017 | 10 days
  The plasma Css,avg of AND017 by multiple administration for 10 consecutive days
Plasma CLss/F of AND017 | 10 days
  The plasma CLss/F of AND017 by multiple administration for 10 consecutive days
Plasma Vss/F of AND017 | 10 days
  The plasma Vss/F of AND017 by multiple administration for 10 consecutive days
Plasma Rac(AUC) of AND017 | 10 days
  The plasma Rac(AUC) of AND017 by multiple administration for 10 consecutive days
Plasma DF of AND017 | 10 days
  The plasma DF of AND017 by multiple administration for 10 consecutive days
PD parameters | 17 days
  Change from baseline levels of EPO
PD parameters | 17 days
  Change from baseline levels of HB
PD parameters | 17 days
  Change from baseline levels of RET

CONTACTS AND LOCATIONS:
Overall Officials: Yusha Zhu, MD PhD, Study Director — Kind Pharmaceuticals LLC
Locations (1):
- Scientia Clinical Research, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No